CLINICAL TRIAL: NCT00050999
Title: A Multicenter Phase III Randomized Double-Blind Placebo-Controlled Study to Evaluate the Efficacy of Two Dose Levels of DAB389IL-2 (9 and 18 Mcg/kg/Day) in Cutaneous T-Cell Lymphoma (CTCL) Patients With Stage Ia-III Disease Who, Following Less Than or Equal to 3 Previous Therapies, Have Recurrent or Persistent Disease That Has Been Biopsy-Documented to Express CD25
Brief Title: Study of ONTAK (Denileukin Diftitox) in Cutaneous T-Cell Lymphoma (CTCL) Patients
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 93-04-11; NCT00002683 (obsolete NCT alias)
Record Dates: First submitted 2002-12-31; First posted 2003-01-03 (Estimated); Last update posted 2008-03-05 (Estimated); Status verified 2008-02

CONDITIONS: Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome
MeSH Terms: conditions — Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome | interventions — denileukin diftitox

INTERVENTIONS:
Drug: ONTAK

SUMMARY:
The purpose of this study is to compare the effectiveness of two dose levels of ONTAK (denileukin diftitox) in treating patients who have recurrent or persistent cutaneous T-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Histopathologically confirmed recurrent or persistent CTCL as determined by reference pathology lab;
* Patient must have had 1 to 3 prior CTCL therapies. Repeated use of the same agent is considered to be 1 therapy unless it is part of a different combination regimen. Only 1 prior combination cytotoxic regimen is permitted. Topical or systemic steroids are not considered a therapy;
* Interleukin-2 receptor (IL-2R) expression on at least 20% of tumor cells as determined by immunohistochemistry.
* Stage IA - III disease and unlikely to progress during the first month on study. Life expectancy of at least 12 months.
* Measurable or evaluable disease. Lymph node involvement no greater than LN2. No CTCL involvement of bone marrow.
* No active CNS disease, kidney or liver disease, significant pulmonary disease, or cardiac disease.
* No systemic infections;
* Willingness to be randomized to a placebo treatment only arm;
* ECOG performance status 0 or 1;

Exclusion Criteria:

• Patients must not have previously received treatment with DAB389IL-2 or DAB486IL 2 (previous candidate compound evaluated in a clinical setting).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 195
Dates: Start 1995-06; Primary Completion 2006-09 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
Objective Rate of Response (ORR), defined as CR + CCR + PR

SECONDARY OUTCOMES:
Time-to-Treatment Failure
Time-to-Progression
Duration of Response

CONTACTS AND LOCATIONS:
Overall Officials: Elyane Lombardy, M.D., Study Director — Ligand Pharmaceuticals
Locations (35):
- University of Texas, M.D. Anderson Cancer Center, Houston, Texas, United States
- Australia (4):
  - Level 4 Department of Haematology Royal North Shore Hospital, Saint Leonard's, New South Wales
  - Westmead Hospital, Department of Haematology, Westmead, New South Wales
  - Mater Misericordiae Adult Hospital, South Brisbane, Queensland
  - Oncology Haematology Radiation Oncology Unit, Princess Alexandra Hospital, Woolloongabba, Queensland
- Austria (2):
  - LKH Universitatsklinikum Graz, Graz
  - Allgemeines Krankenhaus der Stadt Wien, Vienna
- Canada (3):
  - Cross Cancer Centre, Edmonton, Alberta
  - Hamilton Regional Cancer Center, Hamilton, Ontario
  - Jewish General Hospital, Montreal, Quebec
- Germany (8):
  - Universitatsklinikum Charite, Berlin
  - University of Erlangen, Erlangen
  - Universitatsklinikum Essen, Essen
  - J.W. Goethe University Frankfurt, Frankfurt
  - Universitatskrankenhaus Eppendorf, Hamburg
  - Universitatsklinikum Mannheim, Mannheim
  - Universitatsklinikum Munster, Münster
  - Sektion Dermatologische Onkologie, Tübingen
- LUMC, Department of Dermatology, Leiden, Netherlands
- Poland (6):
  - Medical Academy in Gdansk, Dept. of Hematology, Gdansk
  - Regional Oncological Center, Dept. of Chemotherapy, Lodz
  - Klinika Hematoonkologii Akademii Medycznej w Lublinie, Lublin
  - Oddzial Chorob Wewnetrznych i Hematologii, Poznan
  - The Medical University of Warsaw, Central Clinical Hospital, Warsaw
  - Centrum Onkologii-Instytut im. Marii Sklodoskiej-Curie, Warsaw
- Russia (6):
  - Blokhin Russian Cancer Research Center, RAMS, Moscow
  - Burdenko Main Military Clinical Hospital, Moscow
  - Central Research Institute of Skin and Venereal Diseases, Moscow
  - Haematology Research Center RAMS, Moscow
  - St. Petersburg Pavlov State Medical University, Saint Petersburg
  - Samara Regional Clinical Hospital, Samara
- Universitatsspital Zurich Dermatologische Klinik, Zurich, Switzerland
- United Kingdom (3):
  - St. John's Institute of Dermatology, London
  - City Hospital, Nottingham
  - Southampton General Hospital, Southampton

REFERENCES:
- [Derived] Valipour A, Jager M, Wu P, Schmitt J, Bunch C, Weberschock T. Interventions for mycosis fungoides. Cochrane Database Syst Rev. 2020 Jul 7;7(7):CD008946. doi: 10.1002/14651858.CD008946.pub3. PMID 32632956
- [Derived] Duvic M, Geskin L, Prince HM. Duration of response in cutaneous T-cell lymphoma patients treated with denileukin diftitox: results from 3 phase III studies. Clin Lymphoma Myeloma Leuk. 2013 Aug;13(4):377-84. doi: 10.1016/j.clml.2013.02.020. Epub 2013 Jun 14. PMID 23770157